CLINICAL TRIAL: NCT04124289
Title: A Pilot Study to Validate a Functional Pain Scale in Order to Improve the Patient Experience
Brief Title: A Functional Pain Scale to Improve the Patient Experience
Status: Completed | Type: Observational
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 1906-25
Record Dates: First submitted 2019-09-05; First posted 2019-10-11 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pain post surgery: Patients who have completed surgery will be assessed with three types of pain scales. A new pain scale, a functional pain scale (FPS), will be compared to two pain scales that are routinely used: the FACES pain scale and the numeric rating scale (NRS).
  Interventions: Other: Pain measurement using 3 scales

INTERVENTIONS:
Other: Pain measurement using 3 scales — Patients will assess their pain after surgery using three different pain scales.

SUMMARY:
This will be an observational cohort study to evaluate pain measurement after surgery using a new functional pain scale.

DETAILED DESCRIPTION:
Patients admitted for orthopedic surgery may take part in this research. Participants will be assessed using three different pain scales: numeric rating scale (NRS), FACES pain scale and a new functional pain scale (FPS).

ELIGIBILITY:
Inclusion Criteria:

* Completed orthopedic (hip or knee) surgery
* English as primary language and able to read
* Low risk as assessed by Opioid Risk Assessment Tool (ORAT)
* No history of opioid abuse
* Patients with a diagnosis of chronic pain other than the scheduled hip or knee meeting the above criteria may be included.

Exclusion Criteria:

* Previous diagnosis of cognitive impairment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted for orthopedic surgery procedures who will be assessed for pain
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Change in pain score using functional pain scale questionnaire | Through study completion, an average of 4 days.
  Change in pain measurement using new functional pain scale from baseline postoperatively until discharge. The functional pain scale is a scale of 10 descriptive words related to pain and ability to function, ranging from minimal to immobilizing
Change in pain score using FACES pain scale | Through study completion, an average of 4 days.
  Change in pain measurement using FACES pain scale from baseline postoperatively until discharge. The scale includes pictures of facial expressions with correlating numerical scale of 0-10, 0 being no hurt and 10 being the worst hurt.
Change in pain score using numeric 0-10 rating scale | Through study completion, an average of 4 days.
  Change in pain measurement using standard numeric rating scale from baseline postoperatively until discharge. The numeric rating scale is 0-10 where 0 is no pain, 5 is moderate pain and 10 is the worst pain.
Change in functionality | Through study completion, an average of 4 days.
  Change in patient's ability to complete daily functions from baseline postoperatively until discharge. Physical therapy and occupational therapy reports will be reviewed to see if pain appears to interfere with the ability to participate in rehabilitation therapy.

SECONDARY OUTCOMES:
Patient preference for ease of use of the three pain scales (functional, FACES or numerical) | Through study completion, an average of 4 days.
  Questionnaire: Patient will be asked to answer one question to choose which of the three pain scales they prefer for reporting their level of pain. On a scale of 1 to 3 with 1 being the best for reporting pain, the patient will choose which pain scale they would rank a 1.
Provider preference for ease of use of the three pain scales (functional, FACES or numerical) | Through study completion, an average of 4 days.
  Questionnaire: Provider will be asked to answer one question regarding which of the three pain scales they found easiest to complete. On a scale of 1 to 3 with 1 being the best for ease of use, the provider will choose which pain scale they would rank a 1.
Opioid administration | Through study completion, an average of 4 days
  Dose of opioid administered postoperatively during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Harris W Thomas, BSN, RN-BC, Principal Investigator — The Guthrie Clinic
Locations (1):
- Robert Packer Hospital, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No